CLINICAL TRIAL: NCT03540797
Title: The Roles of MDSCs (Myeloid-derived Suppressor Cells) in Adult Patients With Sepsis.
Brief Title: Myeloid-derived Suppressor Cells in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chung Fu-Tsai (Other)
Responsible Party: Sponsor-Investigator, Chung Fu-Tsai, Attending physician, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Other Study IDs: IRB103-6424B
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care unit (ICU) patients with sepsis

SUMMARY:
This study is designed for septic patients, to isolate MDSCs and the correlation of prognosis of sepsis. The purpose of this study hopes to explore the phenomenon and possible mechanisms of MDSCs in patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have known origin of infection .
* Systemic inflammatory response syndrome.

Exclusion Criteria:

* age less than 18 years
* pregnancy
* known anaphylactoid reaction to colloid fluids
* a life expectancy less than 24 hours,
* inability to provide informed, written consent
* Patients receiving nephrotoxic drugs,
* admitted to the hospital following a surgical procedure,
* sepsis more than 72 hours when screening .

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include patients admitted with diagnosis of sepsis in this study.
  Sepsis is defined by the consensus committee of American College of Chest Physicians and Society of Critical Care Medicine. The investigators will interview each patient and their family members, and review the medical records to obtain the baseline information including demographic data, clinical diagnosis, and evidence of dementia or psychiatric disorders. Acute physical and chronic health evaluation (APACHE II) score will be rated by chart review of data obtained within 24 hours of admission. The underlying medical history will also be collected.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival of Intensive care unit (ICU) stay | 28 days

SECONDARY OUTCOMES:
In hospital survival | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Gung Memorial Hospital, Linkou District, Taiwan

IPD SHARING:
Plan to Share IPD: No